CLINICAL TRIAL: NCT05257473
Title: Defining Endpoints in Becker Muscular Dystrophy
Acronym: GRASP-01-002
Status: Active, not recruiting | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Edgewise Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HM20023412; GRASP-BMD (Other: Virginia Commonwealth University)
Record Dates: First submitted 2022-01-25; First posted 2022-02-25 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Becker Muscular Dystrophy; Muscular Dystrophies; Muscular Dystrophy in Children; Muscular Dystrophy, Becker
Keywords: Clinical research; BMD; Becker Muscular Dystrophy; Edgewise Therapeutics
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples will be taken for biomarker development and retained for future research. No clinical diagnosis will be given to patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a 24-month, observational study of 50 participants with Becker muscular dystrophy (BMD)

DETAILED DESCRIPTION:
Becker Muscular Dystrophy (BMD) is most frequently due to in-frame mutations in the dystrophin gene that are associated with reduced levels of frequently shortened dystrophin, though other mutations may be related to the Becker phenotype. There is wide variation in the age of onset and degree of progression, ranging from childhood to late adulthood. The more severe form of dystrophinopathy, Duchenne muscular dystrophy, has a more characteristic rate of progression and overall natural history. The wide variation in severity of progression has led to challenges in the design and conduct of approaching therapeutic trials. There is a need for a more rigorous natural history study to assist in the design of these promising therapeutic trials.

ELIGIBILITY:
Inclusion Criteria:

For ages 6-12

1. Clinically affected (defined as weakness on bedside evaluation in a pattern consistent with BMD)
2. Genetic confirmation of an in-frame dystrophin mutation
3. Ambulatory
4. Willing and able to give informed consent and follow all procedures and requirements

For ages 13 and older

1. Clinically affected (defined as weakness on bedside evaluation in a pattern consistent with BMD)
2. Genetic confirmation of a dystrophin mutation
3. Willing and able to give informed consent and follow all procedures and requirements

For participants in the MRI substudy:

1. Ambulatory, defined as able to walk 10 meters without assistive devices (orthotics allowed)

Exclusion Criteria:

For ages 6-12

1. Out of frame dystrophin mutation
2. Use of chronic corticosteroids at baseline, defined as greater than 6 months of chronic use, will be limited to 20% of the overall population
3. Non-ambulatory, defined as the inability to walk 10 meters without assistive device (excluding orthotics)
4. >16 hours of ventilatory support
5. Any other illness that would interfere with the ability to undergo safe testing or would interfere with interpretation of the results in the opinion of the site investigator.
6. Under the age of 6 at time of enrollment
7. For MR Cohort: Have contraindications to MRI or MRS (e.g., non-MR compatible implanted medical devices or severe claustrophobia)

For ages 13 and older

1. Loss of ambulation prior to age 16
2. Use of chronic corticosteroids, defined as greater than 6 months of chronic use, will be limited to 20% of the overall population
3. Less than 30% of the overall population will be non-ambulatory, defined as the inability to walk 10 meters without assistive device (excluding orthotics)
4. >16 hours of ventilatory support
5. Subjects aged 13-16 only: time to rise >10 seconds
6. For MR Cohort: Have contraindications to MRI or MRS (e.g., non-MR compatible implanted medical devices or severe claustrophobia)

Min Age: 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Becker Muscular Dystrophy affects males.
Study Population: Individuals age 6+ who are clinically affected with Becker Muscular Dystrophy
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-04-13 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
To assess the natural history of measures of muscle function in BMD | Through study completion, an average of 2 years
  North Star Assessment for LGMD (NSAD: The NSAD is a functional scale specifically designed to measure motor performance in individuals with LGMD and is being evaluated in BMD due to the similar limb-girdle pattern of weakness. It consists of 29 items that are considered clinically relevant items from the adapted North Star Ambulatory Assessment and the Motor Function Measure 20 with a maximum score of 54 and higher scores indicate higher functional abilities.
4-Stair Climb | Through study completion, an average of 2 years
  Participants will perform the 4-stair climb with instructions to ascend 4 steps as quickly and as safely possible, using handrails if needed.
100-Meter Timed Test | Through study completion, an average of 2 years
  The participant will be asked to complete 4 laps around 2 cones set 25 meters apart as quickly as safely possible, running if able and the time in seconds is recorded.
PERFORMANCE OF UPPER LIMB 2.0 (PUL) | Through study completion, an average of 2 years
  The PUL is a tool designed for assessing upper limb function in persons with neuromuscular disorders.
HAND HELD DYNAMOMETRY (HHD) AND GRIP | Through study completion, an average of 2 years
  Hand held dynamometry using the MicroFET2 myometer will be utilized to capture isometric strength in target muscle groups. Maximum strength in kilograms will be reported for each muscle group provided a continuous scale variable for analysis. CITEC myometer will be used to measure the and Grip of the subject. These pinch and grip techniques will also capture the maximum strength in newtons for the muscle groups involved.
TIMED UP-AND-GO (TUG) | Through study completion, an average of 2 years
  The TUG will be administered using the appropriate stable seating surface (i.e., cube chair or straight back chair) to achieve 90 degree of both hip and knee flexion when participant is seated with both feet flat on the floor to start. The test should be performed barefoot. The fastest time to stand from the chair, walk 3 meters, and return to seated, will be recorded.
Measures of Pulmonary Function (Seated and supine FVC) | Through study completion, an average of 2 years
  Spirometry will be performed in a sitting and supine position using standardized equipment. Forced vital capacity (FVC) sitting and supine.
Measures of Pulmonary Function (MEP and MIP) | Through study completion, an average of 2 years
  Sitting maximal expiratory and inspiratory pressures (MEP and MIP) will be assessed.
Measures of Pulmonary Function (other) | Through study completion, an average of 2 years
  Use of nocturnal or daytime positive pressure ventilation (PPV) (e.g., BiPAP or CPAP) will be recorded.
Measure of ejection fraction (ECHO) | Through study completion, an average of 2 years
  A transthoracic echocardiogram (ECHO) will be performed. Measures of ejection fraction will be recorded.
Measure of systolic and diastolic function (ECHO) | Through study completion, an average of 2 years
  A transthoracic echocardiogram (ECHO) will be performed. Measures of presence of systolic and diastolic function will be recorded.

OTHER OUTCOMES:
To assess the natural history of MR measures of muscle quality in BMD | Through study completion, an average of 2 years
  MAGNETIC RESONANCE IMAGING FAT FRACTION: This assessment measures fat fraction using chemical shift-based, often called Dixon, imaging and will be performed in axial plane at the thigh and lower leg.
MAGNETIC RESONANCE IMAGING TRANSVERSE RELAXATION TIME (T2) | Through study completion, an average of 2 years
  This assessment measures muscle quality using T2 weighted imaging and will be performed in axial plane at the thigh and lower leg.
MAGNETIC RESONANCE SPECTROSCOPY TRANSVERSE RELAXATION TIME (T2) | Through study completion, an average of 2 years
  Single voxel multiecho magnetic resonance spectra will be acquired for the calculation of water transverse relaxation time.
Biomarker Assessment - Blood Sampling | Through study completion, an average of 2 years
  A blood sample will be collected at the baseline visit to obtain DNA samples for biomarker discovery. Serum will be collected at each in-person visit for other exploratory biomarkers. These samples will be stored in the biorepository, and provide the foundation for future pilot projects, and serve as a resource to the greater BMD community.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas E. Johnson, MD, Principal Investigator — Virginia Commonwealth University
Locations (11):
- United States (9):
  - University of California, Irvine, Orange, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Virginia Commonwealth University, Richmond, Virginia
- University of Auckland, Auckland, New Zealand
- John Walton Muscular Dystrophy Research Centre, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Straub V, Guglieri M. An update on Becker muscular dystrophy. Curr Opin Neurol. 2023 Oct 1;36(5):450-454. doi: 10.1097/WCO.0000000000001191. Epub 2023 Aug 21. PMID 37591308